CLINICAL TRIAL: NCT03084276
Title: Factors That Determine the Responses to Meal Ingestion: Meal Composition
Brief Title: Effect of Meal Composition on the Responses to Meal Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitari Vall d'Hebron Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Other
Other Study IDs: PR(AG)338/2016B
Record Dates: First submitted 2017-03-14; First posted 2017-03-20 (Actual); Last update posted 2017-04-25 (Actual); Status verified 2017-03

CONDITIONS: Healthy
Keywords: meal ingestion; meal composition; postprandial responses; hedonic sensations; homeostatic sensations; new composition

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-fat meal (Experimental)
  Interventions: Other: High-fat meal
- Low-fat meal (Active Comparator)
  Interventions: Other: Low-fat meal

INTERVENTIONS:
Other: High-fat meal — High-fat meal
  Arms: High-fat meal
Other: Low-fat meal — Low-fat meal with the same physical and organoleptic characteristics as the high-calorie meal.
  Arms: Low-fat meal

SUMMARY:
Aim: to determine to what extent meal composition influences postprandial sensations independently of palatability. The postprandial responses to a low-fat (240 Kcal) versus a high-fat (275 Kcal) test meal (150 g humus) with the same physical and organoleptic characteristics (taste, smell, colour, texture, consistency, temperature) will be studied on a cross-over design. The responses to the meals will be tested on 2 different days. Participants (12 non-obese healthy men) will be instructed to eat a standard dinner the day before, to consume a standard breakfast at home after overnight fast, and to report to the laboratory, where the test meal will be administered 3 h after breakfast. Studies will be conducted in a quiet, isolated room with participants sitting on a chair. Perception will be measured at 5 min intervals 10 min before and 20 min after ingestion and at 10 min intervals up to 60 min after the probe meal.

ELIGIBILITY:
Inclusion Criteria:

* non-obese

Exclusion Criteria:

* history of gastrointestinal symptoms
* prior obesity
* use of medications
* history of anosmia and ageusia
* current dieting
* alcohol abuse
* psychological disorders
* eating disorders

Ages: 18 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2017-01-16 (Actual); Primary Completion 2017-03-17 (Actual); Study Completion 2017-03-21 (Actual)

PRIMARY OUTCOMES:
Change in digestive well-being measured after the test meal | 1 day
  Change in average well-being measured by 10 score scales at the end of the test meal.

SECONDARY OUTCOMES:
Change in satiety measured after the test meal | 1 day
  Change in average satiety measured by 10 score scales at the end of the test meal
Change in fullness sensation measured after the test meal | 1 day
  Change in average fullness measured by 10 score scales at the end of the test meal
Change in abdominal discomfort/pain sensation measured after the test meal | 1 day
  Change in average abdominal discomfort/pain measured by 10 score scales at the end of the test meal
Change in mood measured after the test meal | 1 day
  Change in average mood measured by 10 score scales at the end of the test meal.

OTHER OUTCOMES:
Meal palatability | 1 day
  Meal palatability measured by 10 score scales at the end of the test meal.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Vall d'Hebron, Barcelona, Spain